CLINICAL TRIAL: NCT00759304
Title: Evaluation of Aging, Autonomic Nervous System Activity and Cardiovascular Events on a Prospective Cohort of Subjects Aged 65 Years
Brief Title: Evaluation of Aging, Autonomic Nervous System Activity and Cardiovascular Events
Acronym: PROOF
Status: Active, not recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 9808112
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Healthy
Keywords: Aging; cardiovascular risk factors; Autonomic nervous system; stroke; Myocardiac infarction; Neuropsychological evaluation; Prospective cohort
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PROOF cohort: Healthy inhabitants of the city of Saint-Etienne, France, and aged 65 years at the inclusion date.

SUMMARY:
The regulatory effects of the autonomic nervous system (ANS) concern almost all organs which permanently feed information back to this global biological vigilance system controlling allostasis. Heart rate fluctuations are highly dependent on ANS control, making the heart one of the best indicators of ANS activity.

Low ANS activity level is associated with severe cardiac and cerebral events, as well as to death from any cause in the general population.

This PROOF study was hence designed to evaluate ANS activity levels among a healthy retired population, but should these levels decline overtime, to use this as a predictor of cardiovascular and cerebrovascular events, taking into account established cardiovascular risk factors.

DETAILED DESCRIPTION:
The main goal of this PROOF study is to evaluate, on a selected prospective cohort of subjects aged 65 years upon study entry, the prognostic values of ANS activity levels measured at preset times, and more specifically, of its decline over the follow-up period, for fatal and non-fatal cardiovascular and cerebrovascular events.

ELIGIBILITY:
Inclusion Criteria:

* 65 years old
* informed consent signed

Exclusion Criteria:

* prior myocardiac infarction
* prior stroke
* hearth failure
* atrial fibrillation
* insulin-treated diabetes mellitus
* cardiac pacemaker
* disease limiting life expectancy to < 5 years
* contraindication to brain MRI
* living in an institution

Ages: 65 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Subjects were recruited amongst the inhabitants of the city of Saint-Etienne, France, and were eligible if aged 65 at the inclusion date.
Sampling Method: Non-Probability Sample
Enrollment: 1011 (Actual)
Dates: Start 2000-01-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Composite criterion : fatal and non-fatal cardiovascular or cerebrovascular events | During all the study

SECONDARY OUTCOMES:
Presence and severity of clinically silent stroke revealed through brain MRI | Years 1, 3 and 5
Neuropsychological performance | Years 1, 3 and 5
ANS activity measured by heart rate variability + spontaneous baroreflex + blood pressure variability | Years 1, 3 and 5
Biological data : fasting blood glucose, total and HDL cholesterol, triglycerides and CRP | Years 1, 3 and 5

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude BARTHELEMY, MD PhD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- Centre Hospitalier de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roche F, Gaspoz JM, Da Costa A, Isaaz K, Duverney D, Pichot V, Costes F, Lacour JR, Barthelemy JC. Frequent and prolonged asymptomatic episodes of paroxysmal atrial fibrillation revealed by automatic long-term event recorders in patients with a negative 24-hour Holter. Pacing Clin Electrophysiol. 2002 Nov;25(11):1587-93. doi: 10.1046/j.1460-9592.2002.01587.x. PMID 12494616
- [Background] Pichot V, Buffiere S, Gaspoz JM, Costes F, Molliex S, Duverney D, Roche F, Barthelemy JC. Wavelet transform of heart rate variability to assess autonomic nervous system activity does not predict arousal from general anesthesia. Can J Anaesth. 2001 Oct;48(9):859-63. doi: 10.1007/BF03017350. PMID 11606341
- [Result] Barthelemy JC, Pichot V, Dauphinot V, Celle S, Laurent B, Garcin A, Maudoux D, Kerleroux J, Lacour JR, Kossovsky M, Gaspoz JM, Roche F. Autonomic nervous system activity and decline as prognostic indicators of cardiovascular and cerebrovascular events: the 'PROOF' Study. Study design and population sample. Associations with sleep-related breathing disorders: the 'SYNAPSE' Study. Neuroepidemiology. 2007;29(1-2):18-28. doi: 10.1159/000108914. PMID 17898520
- [Result] Gosse P, Roche F, Dauphinot V, Maudoux D, Pichot V, Barthelemy JC. Components of arterial stiffness in a population of 65-year-old subjects: PROOF study. J Hypertens. 2008 Jun;26(6):1138-46. doi: 10.1097/HJH.0b013e3282fa142b. PMID 18475151
- [Result] Rouch I, Anterion CT, Dauphinot V, Kerleroux J, Roche F, Barthelemy JC, Laurent B. Cognitive complaints, neuropsychological performance and affective disorders in elderly community residents. Disabil Rehabil. 2008;30(23):1794-802. doi: 10.1080/09638280701667825. PMID 18608410
- [Derived] Vogrig M, Berger AE, Bourlet T, Waeckel L, Haccourt A, Chanavat A, Hupin D, Roche F, Botelho-Nevers E, Pozzetto B, Paul S. Monitoring of Both Humoral and Cellular Immunities Could Early Predict COVID-19 Vaccine Efficacy Against the Different SARS-CoV2 Variants. J Clin Immunol. 2023 Jan;43(1):31-45. doi: 10.1007/s10875-022-01354-x. Epub 2022 Aug 25. PMID 36006568
- [Derived] Hupin D, Raffin J, Barth N, Berger M, Garet M, Stampone K, Celle S, Pichot V, Bongue B, Barthelemy JC, Roche F. Even a Previous Light-Active Physical Activity at Work Still Reduces Late Myocardial Infarction and Stroke in Retired Adults Aged>65 Years by 32%: The PROOF Cohort Study. Front Public Health. 2019 Mar 19;7:51. doi: 10.3389/fpubh.2019.00051. eCollection 2019. PMID 30941340
- [Derived] Sforza E, Millasseau S, Hupin D, Barthelemy JC, Roche F. Arterial stiffness alteration and obstructive sleep apnea in an elderly cohort free of cardiovascular event history: the PROOF cohort study. Sleep Breath. 2019 Mar;23(1):201-208. doi: 10.1007/s11325-018-1683-x. Epub 2018 Jun 26. PMID 29946946
- [Derived] Celle S, Boutet C, Annweiler C, Barthelemy JC, Roche F. Sleep apnoea in the asymptomatic elderly: a real issue for the brain? Eur Respir J. 2018 Jun 14;51(6):1702450. doi: 10.1183/13993003.02450-2017. Print 2018 Jun. PMID 29903827
- [Derived] Monneret D, Barthelemy JC, Hupin D, Maudoux D, Celle S, Sforza E, Roche F. Serum lipid profile, sleep-disordered breathing and blood pressure in the elderly: a 10-year follow-up of the PROOF-SYNAPSE cohort. Sleep Med. 2017 Nov;39:14-22. doi: 10.1016/j.sleep.2017.07.028. Epub 2017 Sep 18. PMID 29157582
- [Derived] Saint Martin M, Labeix P, Garet M, Thomas T, Barthelemy JC, Collet P, Roche F, Sforza E. Does Subjective Sleep Affect Bone Mineral Density in Older People with Minimal Health Disorders? The PROOF Cohort. J Clin Sleep Med. 2016 Nov 15;12(11):1461-1469. doi: 10.5664/jcsm.6266. PMID 27655463
- [Derived] Sforza E, Saint Martin M, Thomas T, Collet P, Garet M, Barthelemy JC, Roche F. Risk factors of osteoporosis in healthy elderly with unrecognized obstructive sleep apnea: role of physical activity. Sleep Med. 2016 Jun;22:25-32. doi: 10.1016/j.sleep.2016.04.010. Epub 2016 Jun 7. PMID 27544832
- [Derived] Sforza E, Saint Martin M, Barthelemy JC, Roche F. Mood disorders in healthy elderly with obstructive sleep apnea: a gender effect. Sleep Med. 2016 Mar;19:57-62. doi: 10.1016/j.sleep.2015.11.007. Epub 2015 Nov 25. PMID 27198948
- [Derived] Boutet C, Vassal F, Celle S, Schneider FC, Barthelemy JC, Laurent B, Barral FG, Roche F. Incidental findings on brain magnetic resonance imaging in the elderly:the PROOF study. Brain Imaging Behav. 2017 Feb;11(1):293-299. doi: 10.1007/s11682-016-9519-4. PMID 26843003
- [Derived] Sforza E, Celle S, Saint-Martin M, Barthelemy JC, Roche F. Hippocampus volume and subjective sleepiness in older people with sleep-disordered breathing: a preliminary report. J Sleep Res. 2016 Apr;25(2):190-3. doi: 10.1111/jsr.12367. Epub 2015 Dec 14. PMID 26662175
- [Derived] Sforza E, Pichot V, Martin MS, Barthelemy JC, Roche F. Prevalence and determinants of subjective sleepiness in healthy elderly with unrecognized obstructive sleep apnea. Sleep Med. 2015 Aug;16(8):981-6. doi: 10.1016/j.sleep.2015.03.010. Epub 2015 Apr 15. PMID 26141008
- [Derived] Sforza E, Sabri M, DaCosta A, Isaaz K, Barthelemy JC, Roche F. Echocardiographic Findings in Healthy Elderly People with Unrecognized Sleep Disordered Breathing. J Clin Sleep Med. 2015 Sep 15;11(9):975-80. doi: 10.5664/jcsm.5006. PMID 25902826
- [Derived] Saint Martin M, Roche F, Thomas-Anterion C, Barthelemy JC, Sforza E; PROgnostic OF cardiovascular and cerebrovascular events study group. Eight-year parallel change in baroreflex sensitivity and memory function in a sample of healthy older adults. J Am Geriatr Soc. 2015 Feb;63(2):270-5. doi: 10.1111/jgs.13252. Epub 2015 Feb 2. PMID 25641086
- [Derived] Martin MS, Sforza E, Roche F, Barthelemy JC, Thomas-Anterion C; PROOF study group. Sleep breathing disorders and cognitive function in the elderly: an 8-year follow-up study. the proof-synapse cohort. Sleep. 2015 Feb 1;38(2):179-87. doi: 10.5665/sleep.4392. PMID 25325480
- [Derived] Sforza E, Saint Martin M, Barthelemy JC, Roche F. Association of self-reported sleep and hypertension in non-insomniac elderly subjects. J Clin Sleep Med. 2014 Sep 15;10(9):965-71. doi: 10.5664/jcsm.4026. PMID 25142770
- [Derived] Saint Martin M, Sforza E, Thomas-Anterion C, Barthelemy JC, Roche F; PROOF Study Group. Baroreflex sensitivity, vascular risk factors, and cognitive function in a healthy elderly population: the PROOF cohort. J Am Geriatr Soc. 2013 Dec;61(12):2096-2102. doi: 10.1111/jgs.12548. Epub 2013 Nov 26. PMID 24279643
- [Derived] Sforza E, Thomas T, Barthelemy JC, Collet P, Roche F. Obstructive sleep apnea is associated with preserved bone mineral density in healthy elderly subjects. Sleep. 2013 Oct 1;36(10):1509-15. doi: 10.5665/sleep.3046. PMID 24082310
- [Derived] Martin MS, Sforza E, Barthelemy JC, Thomas-Anterion C, Roche F. Sleep perception in non-insomniac healthy elderly: a 3-year longitudinal study. Rejuvenation Res. 2014 Feb;17(1):11-8. doi: 10.1089/rej.2013.1457. PMID 24033249
- [Derived] Chouchou F, Pichot V, Pepin JL, Tamisier R, Celle S, Maudoux D, Garcin A, Levy P, Barthelemy JC, Roche F; PROOF Study Group. Sympathetic overactivity due to sleep fragmentation is associated with elevated diurnal systolic blood pressure in healthy elderly subjects: the PROOF-SYNAPSE study. Eur Heart J. 2013 Jul;34(28):2122-31, 2131a. doi: 10.1093/eurheartj/eht208. Epub 2013 Jun 11. PMID 23756334
- [Derived] Degache F, Sforza E, Dauphinot V, Celle S, Garcin A, Collet P, Pichot V, Barthelemy JC, Roche F; PROOF Study Group. Relation of central fat mass to obstructive sleep apnea in the elderly. Sleep. 2013 Apr 1;36(4):501-7. doi: 10.5665/sleep.2532. PMID 23564997
- [Derived] Dauphinot V, Rouch I, Kossovsky MP, Pichot V, Dorey JM, Krolak-Salmon P, Laurent B, Roche F, Barthelemy JC. Depressive symptoms and autonomic nervous system dysfunction in an elderly population-based study: the PROOF study. J Affect Disord. 2012 Dec 20;143(1-3):153-9. doi: 10.1016/j.jad.2012.05.045. Epub 2012 Aug 19. PMID 22910448
- [Derived] Sforza E, Gauthier M, Crawford-Achour E, Pichot V, Maudoux D, Barthelemy JC, Roche F. A 3-year longitudinal study of sleep disordered breathing in the elderly. Eur Respir J. 2012 Sep;40(3):665-72. doi: 10.1183/09031936.00133011. Epub 2012 Mar 9. PMID 22408210
- [Derived] Tonnesen P, Lauri H, Perfekt R, Mann K, Batra A. Efficacy of a nicotine mouth spray in smoking cessation: a randomised, double-blind trial. Eur Respir J. 2012 Sep;40(3):548-54. doi: 10.1183/09031936.00155811. Epub 2012 Feb 9. PMID 22323576
- [Derived] Assoumou HG, Bertholon F, Barthelemy JC, Pichot V, Celle S, Gosse P, Gaspoz JM, Roche F. Alteration of baroreflex sensitivity in the elderly: the relationship with metabolic syndrome components. Int J Cardiol. 2012 Mar 8;155(2):333-5. doi: 10.1016/j.ijcard.2011.12.050. Epub 2012 Jan 10. No abstract available. PMID 22240751
- [Derived] Sforza E, Chouchou F, Pichot V, Barthelemy JC, Roche F. Heart rate increment in the diagnosis of obstructive sleep apnoea in an older population. Sleep Med. 2012 Jan;13(1):21-8. doi: 10.1016/j.sleep.2011.04.011. Epub 2011 Nov 21. PMID 22104544
- [Derived] Dauphinot V, Barthelemy JC, Pichot V, Celle S, Sforza E, Achour-Crawford E, Gosse P, Roche F. Autonomic activation during sleep and new-onset ambulatory hypertension in the elderly. Int J Cardiol. 2012 Feb 23;155(1):155-9. doi: 10.1016/j.ijcard.2011.10.097. Epub 2011 Nov 9. PMID 22078984
- [Derived] Ntougou Assoumou HG, Pichot V, Barthelemy JC, Dauphinot V, Celle S, Collet P, Gaspoz JM, Roche F. Obesity-related autonomic nervous system disorders are best associated with body fat mass index, a new indicator. Int J Cardiol. 2011 Nov 17;153(1):111-3. doi: 10.1016/j.ijcard.2011.09.031. Epub 2011 Oct 2. No abstract available. PMID 21963211
- [Derived] Chouchou F, Sforza E, Celle S, Pichot V, Maudoux D, Garcin A, Barthelemy JC, Roche F; PROOF Study Group. Pulse transit time in screening sleep disordered breathing in an elderly population: the PROOF-SYNAPSE study. Sleep. 2011 Aug 1;34(8):1051-9. doi: 10.5665/SLEEP.1160. PMID 21804667
- [Derived] Castro-Lionard K, Thomas-Anterion C, Crawford-Achour E, Rouch I, Trombert-Paviot B, Barthelemy JC, Laurent B, Roche F, Gonthier R. Can maintaining cognitive function at 65 years old predict successful ageing 6 years later? The PROOF study. Age Ageing. 2011 Mar;40(2):259-65. doi: 10.1093/ageing/afq174. Epub 2011 Jan 20. PMID 21252039
- [Derived] Sforza E, Chouchou F, Collet P, Pichot V, Barthelemy JC, Roche F. Sex differences in obstructive sleep apnoea in an elderly French population. Eur Respir J. 2011 May;37(5):1137-43. doi: 10.1183/09031936.00043210. Epub 2010 Sep 3. PMID 20817711